CLINICAL TRIAL: NCT02371213
Title: Antenatal Care Health Education Intervened by Social Networking on Mobile Phone Compared With Usual Care to Improve Maternal and Neonatal Outcomes: Randomized Controlled Trial
Brief Title: Social Networking on Mobile Phone to Improve Maternal and Neonatal Outcomes
Acronym: HISONET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nopparatrajathanee Hospital (Other)
Responsible Party: Principal Investigator, Krissada Tomyabatra, Dr, Nopparatrajathanee Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HISONET-1
Record Dates: First submitted 2015-02-19; First posted 2015-02-25 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Premature Birth
Keywords: Social Networking; Mobile phone; Antenatal Care; Health education; Maternal outcome; Neonatal outcome
MeSH Terms: conditions — Premature Birth; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- social networking on mobile phone (Experimental): Audio-video media via social networking on mobile phone to antenatal women from the first ANC visit four times every month and four times biweekly plus usual antenatal care group-health education
  Interventions: Other: social networking on mobile phone
- no social networking on mobile phone (No Intervention): usual antenatal care group-health education

INTERVENTIONS:
Other: social networking on mobile phone — Audio-video media about serious complications such as labor pain, vaginal bleeding, water breaking and fewer fetal movement via social networking application on mobile phone to antenatal women from the first ANC visit four times every month and four times biweekly
  Arms: social networking on mobile phone

SUMMARY:
The purpose of the study is to determine whether social networking on mobile phone in antenatal care health education is effective in the improvement of maternal and neonatal outcomes compared with usual antenatal care.

DETAILED DESCRIPTION:
Health Education Intervention with Social Networking (HISONET) is a open-label randomized controlled trial. The objective of this study is to determine the efficacy of social networking media on mobile phone intervention in antenatal care (ANC) group-health education compared with usual ANC health education. The incidence of preterm delivery and major neonatal morbidity including respiratory distress syndrome, stillbirth and perinatal mortality in women delivering from 28 to 36 weeks' gestation are significant outcomes in a randomized prospective design. Preterm delivery occurs in approximately 9.6% as global incidence, and about 11.1% in South-Eastern Asia. Forty-four percent of child under 5 years died in neonatal period. Preterm birth is one of the three leading causes of neonatal death which 15% died from preterm birth complications such as respiratory distress syndrome, intraventricular hemorrhage, necrotizing entercolitis, and sepsis. Recent studies demonstrate that Short Message Service (SMS) on mobile phone intervention in antenatal care can increase numbers of ANC attendance to WHO recommendation of four or more visits and decrease in perinatal mortality.

Social networking on mobile phone has been increasingly used in daily life of both healthcare personnel and women who attend ANC clinic. However, there is lack of evidence that demonstrates the effect of social networking on mobile phone to improve maternal and neonatal outcomes. LINE, a mobile application, is a popular one of many social networking applications. So, health education through LINE of antenatal women about serious complications such as labor pain, bleeding, water breaking and fewer fetal movement during pregnancy may encourage them to come to the hospital as early as possible. Early diagnosis of premature labor provides early management and better maternal and neonatal outcomes. So, a randomized controlled trial should be conducted to answer these questions.

ELIGIBILITY:
Inclusion Criteria:

* women who attend antenatal care clinic and have intention to deliver at the study hospital.
* Thai race
* participant or husband or relatives is an owner of mobile phone with social networking application

Exclusion Criteria:

* participant is known by other one in different study arm (contamination)
* cannot be assess on wel-being about privacy, delivery failure and misinterpretation of media via social network after complete study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1160 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Rate of Premature birth | before 37 weeks gestation
  Preterm is defined as babies born alive before 37 weeks of pregnancy are completed [WHO]

SECONDARY OUTCOMES:
Rate of Respiratory Distress Syndrome | 28 days after birth
  Respiratory distress syndrome (RDS) is a breathing disorder that affects newborns [NIH]
Rate of Stillbirth | after 28 weeks' gestation to birth
  A baby born with no signs of life at or after 28 weeks' gestation [WHO]
Rate of Perinatal Mortality | after 28 weeks' gestation to the first week of life [WHO]
  Perinatal mortality refers to the number of stillbirths and deaths in the first week of life (early neonatal mortality). [WHO]

CONTACTS AND LOCATIONS:
Overall Officials: Krissada Tomyabatra, MD, RTCOG, Principal Investigator — Nopparatrajathanee Hospital
Locations (1):
- Nopparatrajathanee Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu L, Oza S, Hogan D, Perin J, Rudan I, Lawn JE, Cousens S, Mathers C, Black RE. Global, regional, and national causes of child mortality in 2000-13, with projections to inform post-2015 priorities: an updated systematic analysis. Lancet. 2015 Jan 31;385(9966):430-40. doi: 10.1016/S0140-6736(14)61698-6. Epub 2014 Sep 30. PMID 25280870
- [Background] Beck S, Wojdyla D, Say L, Betran AP, Merialdi M, Requejo JH, Rubens C, Menon R, Van Look PF. The worldwide incidence of preterm birth: a systematic review of maternal mortality and morbidity. Bull World Health Organ. 2010 Jan;88(1):31-8. doi: 10.2471/BLT.08.062554. Epub 2009 Sep 25. PMID 20428351
- [Background] Jareethum R, Titapant V, Chantra T, Sommai V, Chuenwattana P, Jirawan C. Satisfaction of healthy pregnant women receiving short message service via mobile phone for prenatal support: A randomized controlled trial. J Med Assoc Thai. 2008 Apr;91(4):458-63. PMID 18556852
- [Background] Lund S, Hemed M, Nielsen BB, Said A, Said K, Makungu MH, Rasch V. Mobile phones as a health communication tool to improve skilled attendance at delivery in Zanzibar: a cluster-randomised controlled trial. BJOG. 2012 Sep;119(10):1256-64. doi: 10.1111/j.1471-0528.2012.03413.x. Epub 2012 Jul 17. PMID 22805598
- [Background] Lund S, Nielsen BB, Hemed M, Boas IM, Said A, Said K, Makungu MH, Rasch V. Mobile phones improve antenatal care attendance in Zanzibar: a cluster randomized controlled trial. BMC Pregnancy Childbirth. 2014 Jan 17;14:29. doi: 10.1186/1471-2393-14-29. PMID 24438517
- [Background] Lund S, Rasch V, Hemed M, Boas IM, Said A, Said K, Makundu MH, Nielsen BB. Mobile phone intervention reduces perinatal mortality in zanzibar: secondary outcomes of a cluster randomized controlled trial. JMIR Mhealth Uhealth. 2014 Mar 26;2(1):e15. doi: 10.2196/mhealth.2941. PMID 25098184
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276